CLINICAL TRIAL: NCT04913727
Title: Prediction of Reverse Remodeling and Outcome in Patients With Severe Secondary Mitral Valve Regurgitation Undergoing Transcatheter Edge-to-edge Mitral Valve Repair
Acronym: PRE-MITRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Cardiocentro Ticino (Other); Triemli Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-00704
Record Dates: First submitted 2021-05-27; First posted 2021-06-04 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Severe Mitral Regurgitation
Keywords: Cardiac magnet resonance (CMR); Mitral Regurgitation; Transcatheter mitral edge-to-edge repair; MitraClip; CMR feature tracking; Parametric mapping
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients undergoing transcatheter mitral edge-to-edge repair in this single-arm study.
  Interventions: Diagnostic Test: Cardiac magnetic resonance imaging before the procedure; Procedure: Transcatheter mitral edge-to-edge repair.

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance imaging before the procedure — CMR image acquisition with previously mentioned analysis
Procedure: Transcatheter mitral edge-to-edge repair. — Included patients will undergo Transcatheter mitral edge-to-edge repair.

SUMMARY:
The investigators' hypothesis is that CMR tissue characterization and myocardial function analysis acquired by CMR feature tracking technique predict reverse remodeling in patients with severe secondary mitral regurgitation (MR) undergoing transcatheter mitral edge-to-edge repair.

DETAILED DESCRIPTION:
Diametrically opposed results of the COAPT- and the MITRA-FR trial have demonstrated the need for additional evidence in the field of transcatheter mitral edge-to-edge repair. Reverse left ventricular remodeling after treatment of severe secondary mitral regurgitation can indicate treatment response and is associated with positive outcomes.

However, so far it is reverse remodeling, respectively treatment response is difficult to predict, which complicates patient selection for mitral edge-to-edge repair. Previous studies have shown, that focal (late gadolinium enhancement (LGE)) but not diffuse myocardial fibrosis (T1 mapping and extracellular volume fraction (ECV)) burden quantification using CMR predicts reverse left ventricular remodeling following cardiac resynchronization therapy in patients with heart failure with reduced ejection fraction (HFrEF). On the other hand, myocardial T1 mapping was predictive for beneficial left ventricular remodeling after long-term heart failure therapy. Furthermore, in patients with HFrEF, LGE is associated with clinical outcome and an incremental predictive value to left ventricular dimensions and function. However, as only 1/3 of HFrEF patients show LGE, subtle fibrosis might be missed. Recently the investigators have shown that different novel fibrosis detection techniques (naive T1 mapping, mean ECV and λGd being the delta of pre- and post T1 mapping and ECV calculation) all demonstrated strong association with outcome in patients with heart failure.

The investigators' hypothesis is that these markers (CMR tissue characterization and myocardial function analysis acquired by a CMR feature tracking) might also be helpful in predicting reverse remodeling after transcatheter mitral edge-to-edge repair. This project might help to understand the pathophysiology of the disease in patients with secondary mitral regurgitation, improve risk stratification in this clinical setting, and optimize selection of patients who benefit from transcatheter mitral edge-to-edge repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe secondary MR characterized, according to the European guidelines and recommendations, by a regurgitant volume ≥30 mL/beat or an effective regurgitant orifice ≥20 mm².
* Symptomatic patients with New York Heart Association Class ≥II.
* Left ventricular ejection fraction between 15% and 50%.
* Optimal standard of care therapy for heart failure according to investigator.
* Not eligible for a mitral surgery intervention according to the Heart Team.
* Patients who have the ability to understand the requirements of the study and provide written consent/assent to participate and agree to abide by the study requirements.

Exclusion Criteria:

* Participants younger than 18 years
* Pregnancy or breastfeeding
* Severe impaired renal function (GFR < 15 ml/min)
* Patients with untreated severe concomitant valve disease (e.g. severe tricuspid valve regurgitation, aortic stenosis)
* The patient has a medical condition, serious concurrent illness, or extenuating circumstance that would significantly decrease study compliance, including all prescribed follow-up
* The patient has contraindications to CMR, including: Implanted non-CMR conditional metallic implants, pacemaker, intracardiac defibrillator, neurostimulator, epicardial pacemaker leads, or any abandoned leads, ferromagnetic aneurysm clip, ferromagnetic halo device, cochlear implants, implanted infusion pumps or severe claustrophobia
* The patient is clinically unstable or has stage D congestive heart failure or inability to lay flat for 60 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with reverse remodeling after 12 months | 12 months after mitral edge-to-edge repair
  Defined as ≥10% reduction in left ventricular end-diastolic volume in patients with successful MR reduction to grade 2+ or less 12 months after mitral edge-to-edge repair assessed by echocardiography.

SECONDARY OUTCOMES:
Rate of patients with procedural and device success | 24 months after mitral edge-to-edge repair
  Procedural and device success as defined according to the criteria of the Mitral Valve Academic Research Consortium
Rate of patients with reverse remodeling after 6 and 24 months | 6 and 24 months after mitral edge-to-edge repair
  Reverse remodeling at 6 and 24 months, defined according to previously mentioned criteria.
Change of left ventricular sphericity index | 6, 12 and 24 months after mitral edge-to-edge repair
  Echocardiographic assessment of LV sphericity index measured using the LV short/long axis dimension ratio in the end-diastolic four-chamber apical view.
Change in NT-proBNP levels | 6, 12 and 24 months after mitral edge-to-edge repair
  Change in NT-proBNP levels as an indirect sign of changes in left ventricular filling pressure, fibrosis and reverse remodeling will be measured in clinically indicated follow-ups at different time points after the intervention.
All cause death | 6, 12 and 24 months after mitral edge-to-edge repair
  Occurence of death from any cause
Cardiovascular death | 6, 12 and 24 months after mitral edge-to-edge repair
  Occurence of death from cardiovascular reason
Rate of patients with heart-failure related hospitalization | 6, 12 and 24 months after mitral edge-to-edge repair
  Hospitalizations for heart failure within the observation time will be systematically recorded.
Change in NYHA class | 6, 12 and 24 months after mitral edge-to-edge repair
  Change in NYHA class ≥ +/- 1 compared to baseline NYHA-class before mitral edge-to-edge repair.
Change in myocardial strain | Within 24 months after mitral edge-to-edge repair
  Clinically indicated follow-up imaging (CMR) will be analyzed by CMR feature tracking
Change in left ventricular ejection fraction | 6, 12 and 24 months after mitral edge-to-edge repair
  Echocardiographic assessment of left ventricular ejection fraction measured according to biplane Simpson disk summation method.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph MD Gräni, PHD, Principal Investigator — Department of Cardiology, University Hospital Bern, Inselspital, Bern
Locations (1):
- Department of Cardiology, University Hospital Bern, Inselspital, Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stone GW, Lindenfeld J, Abraham WT, Kar S, Lim DS, Mishell JM, Whisenant B, Grayburn PA, Rinaldi M, Kapadia SR, Rajagopal V, Sarembock IJ, Brieke A, Marx SO, Cohen DJ, Weissman NJ, Mack MJ; COAPT Investigators. Transcatheter Mitral-Valve Repair in Patients with Heart Failure. N Engl J Med. 2018 Dec 13;379(24):2307-2318. doi: 10.1056/NEJMoa1806640. Epub 2018 Sep 23. PMID 30280640
- [Result] Obadia JF, Messika-Zeitoun D, Leurent G, Iung B, Bonnet G, Piriou N, Lefevre T, Piot C, Rouleau F, Carrie D, Nejjari M, Ohlmann P, Leclercq F, Saint Etienne C, Teiger E, Leroux L, Karam N, Michel N, Gilard M, Donal E, Trochu JN, Cormier B, Armoiry X, Boutitie F, Maucort-Boulch D, Barnel C, Samson G, Guerin P, Vahanian A, Mewton N; MITRA-FR Investigators. Percutaneous Repair or Medical Treatment for Secondary Mitral Regurgitation. N Engl J Med. 2018 Dec 13;379(24):2297-2306. doi: 10.1056/NEJMoa1805374. Epub 2018 Aug 27. PMID 30145927
- [Result] Praz F, Grasso C, Taramasso M, Baumbach A, Piazza N, Tamburino C, Windecker S, Maisano F, Prendergast B. Mitral regurgitation in heart failure: time for a rethink. Eur Heart J. 2019 Jul 14;40(27):2189-2193. doi: 10.1093/eurheartj/ehz222. No abstract available. PMID 31005977
- [Result] Grani C, Eichhorn C, Biere L, Murthy VL, Agarwal V, Kaneko K, Cuddy S, Aghayev A, Steigner M, Blankstein R, Jerosch-Herold M, Kwong RY. Prognostic Value of Cardiac Magnetic Resonance Tissue Characterization in Risk Stratifying Patients With Suspected Myocarditis. J Am Coll Cardiol. 2017 Oct 17;70(16):1964-1976. doi: 10.1016/j.jacc.2017.08.050. PMID 29025553
- [Result] Grani C, Biere L, Eichhorn C, Kaneko K, Agarwal V, Aghayev A, Steigner M, Blankstein R, Jerosch-Herold M, Kwong RY. Incremental value of extracellular volume assessment by cardiovascular magnetic resonance imaging in risk stratifying patients with suspected myocarditis. Int J Cardiovasc Imaging. 2019 Jun;35(6):1067-1078. doi: 10.1007/s10554-019-01552-6. Epub 2019 Feb 12. PMID 30756221
- [Result] Grani C, Eichhorn C, Biere L, Kaneko K, Murthy VL, Agarwal V, Aghayev A, Steigner M, Blankstein R, Jerosch-Herold M, Kwong RY. Comparison of myocardial fibrosis quantification methods by cardiovascular magnetic resonance imaging for risk stratification of patients with suspected myocarditis. J Cardiovasc Magn Reson. 2019 Feb 28;21(1):14. doi: 10.1186/s12968-019-0520-0. PMID 30813942